CLINICAL TRIAL: NCT07327060
Title: Effect of Intraoral Camera-Assisted Parent Training on Children's Oral Hygiene and Parent Oral Health Literacy: A Randomized Controlled Trial
Brief Title: Intraoral Camera-Assisted Parent Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Melis AKYILDIZ, assistant prof, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mgungor
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Oral Health Literacy; Oral Health Care; Intraoral Images; Periodontal Index; Gingival Index; Caries
Keywords: Oral health literacy; Oral Health Care; İntraoral camera

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, controlled, parallel-group design. Participants are randomly assigned to the intervention or control group using computer-based block randomization through Random.Org (Randomness and Integrity Services Ltd., Ireland) to ensure fair and concealed allocation. Both groups are followed during the same period. Because the intervention is educational, blinding of participants and educators is not possible; however, outcome assessors are blinded to reduce bias. This design helps us evaluate whether intraoral camera-assisted education, in addition to standard oral hygiene instruction, improves children's oral health outcomes and increases parents' oral health literacy.
Who Masked: Outcomes Assessor
Masking Description: For both children and parents, the intraoral camera-assisted education or verbal instruction will be applied clearly within each group, and parents will be informed about the procedures and the study plan. To increase the scientific validity and reliability of the results, oral examinations and data collection will be done by different people. In this way, the assessors will stay blinded to the participants' group allocation during all evaluations, ensuring that the data collected are objective. The same blinding will be used for the Occlusal Plaque Index (OPI) assessment, so the examiner will evaluate plaque on first permanent molars without knowing whether the child received intraoral camera-assisted education or standard verbal instruction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoral Camera-Assisted Oral Hygiene Education (Experimental): In the intervention group, explanations provided during the oral examination will be visualized using an intraoral camera. After recording oral hygiene scores, a disclosing agent will be applied to the teeth. Following gentle rinsing and isolation, areas stained by plaque and not effectively cleaned will be highlighted, and brushing will be demonstrated accordingly. Using the Modified Stillman technique, the specific areas requiring toothbrush contact will be shown directly in the patient's mouth with intraoral camera visualization. Signs of gingival inflammation such as redness or swelling, as well as caries and plaque deposits, will also be displayed in real time. This approach individualizes the education, enabling both the child and parent to better understand and retain the oral hygiene instructions.
  Interventions: Behavioral: Intraoral Camera-Assisted Oral Hygiene Education; Device: Intraoral Photography of Permanent First Molars; Behavioral: Turkish Version of the Oral Health Literacy Assessment Task for Pediatric Dentistry (TOHLAT-P); Other: Parent and Child Satisfaction Survey
- Standard Verbal Oral Hygiene Education (Active Comparator): Children in the control group undergo oral examination at the dental unit using a mirror and probe. Standard verbal oral hygiene education is provided to children and parents, including information on dental plaque, oral hygiene importance, and treatment needs. Brushing is demonstrated on a model using the Modified Stillman technique to ensure effective plaque control without harming the gingiva. For partially erupted permanent first molars, the "cross brushing" technique with horizontal bucco-lingual movements is also explained.
  Interventions: Behavioral: Standard Verbal Oral Hygiene Education; Device: Intraoral Photography of Permanent First Molars; Behavioral: Turkish Version of the Oral Health Literacy Assessment Task for Pediatric Dentistry (TOHLAT-P)

INTERVENTIONS:
Behavioral: Intraoral Camera-Assisted Oral Hygiene Education — Participants receive individualized oral hygiene education using an intraoral camera. Dental findings such as plaque, caries, and gingival inflammation are visualized in real time. Disclosing agents highlight plaque-covered areas, and brushing demonstrations are performed directly on the child's teeth using the Modified Stillman and cross-brushing techniques. Parents and children receive visual feedback to reinforce proper oral hygiene practices.
  Arms: Intraoral Camera-Assisted Oral Hygiene Education
Behavioral: Standard Verbal Oral Hygiene Education — Participants receive standard verbal oral hygiene education using a brushing model. The Modified Stillman and cross-brushing techniques are demonstrated verbally and on the model. Oral hygiene principles, plaque control, and the importance of regular brushing are explained to both children and parents.
  Arms: Standard Verbal Oral Hygiene Education
Device: Intraoral Photography of Permanent First Molars — Occlusal surfaces of permanent first molars will be photographed using the EZCAM VATECH intraoral camera to document plaque accumulation. The photographs will be shown only to participants in the camera-assisted education group during oral hygiene instruction. These images will help them see plaque areas and understand correct brushing. The control group will receive only verbal education and will not view the photographs. All images will be stored securely and used only for evaluation in the study.
Behavioral: Turkish Version of the Oral Health Literacy Assessment Task for Pediatric Dentistry (TOHLAT-P) — Parental oral health literacy, knowledge about preventive dental care, and their ability to help their child with oral hygiene will be measured using the Turkish version of the Oral Health Literacy Assessment Task for Pediatric Dentistry (TOHLAT-P). This tool evaluates parents' understanding and use of oral health information. Higher scores indicate better oral health literacy.
Other: Parent and Child Satisfaction Survey — A structured questionnaire was given to children and parents in the intraoral camera education group. The aim was to evaluate their satisfaction with the education process. The questionnaire focused on the usability of the intraoral camera and how helpful it was during dental education.
  Arms: Intraoral Camera-Assisted Oral Hygiene Education

SUMMARY:
The aim of this randomized controlled trial is to test the null hypothesis that parent education using an intraoral camera has no effect on children's oral hygiene levels, parental oral health literacy, or plaque accumulation on first permanent molars compared with standard verbal education. 40 children aged 5-7 and their parents will be randomly assigned to two groups. The intervention group will receive real-time visualization of dental conditions and brushing techniques using an intraoral camera, while the control group will receive standard verbal education using a brushing model. Outcomes include children's plaque and gum health and ICDAS caries scores. Secondary outcomes include Occlusal Plaque Index (OPI) on first molars. Assessments will be conducted at baseline and 1-month follow-up. This study tests whether intraoral camera-assisted education leads to better oral hygiene outcomes in children, improves parents' oral health literacy, and reduces plaque accumulation on the first permanent molars compared to standard verbal education.

DETAILED DESCRIPTION:
Dental caries is a common problem in children, and teaching good oral hygiene is important for prevention. Parents play a key role in protecting their children's teeth, especially when the first permanent molars erupt, because these teeth are more sensitive to plaque and caries. In pediatric dentistry, it is known that when parents have better oral health literacy, their children tend to show better oral health outcomes, making parental literacy an important factor.

Because of this, education methods that allow parents and children to see the mouth clearly may be more effective. Using an intraoral camera provides real-time visual feedback, so children and parents can directly observe plaque, caries, and brushing mistakes. This may increase motivation, support correct brushing techniques, and improve parents' understanding of oral health.

The aim of this study is to determine whether intraoral camera-assisted education can improve children's oral hygiene and increase parents' oral health awareness and literacy more than standard verbal education.

Based on this aim, the study tested the following hypotheses:

Null Hypothesis (H0a): Intraoral camera-assisted education has no effect on improving children's oral hygiene levels.

Alternative Hypothesis (H1a): Intraoral camera-assisted education improves children's oral hygiene levels.

Null Hypothesis (H0b): Intraoral camera-assisted education has no effect on improving parental oral health literacy.

Alternative Hypothesis (H1b): Intraoral camera-assisted education improves parental oral health literacy.

Null Hypothesis (H0c): Intraoral camera-assisted education has no effect on plaque accumulation on first permanent molars.

Alternative Hypothesis (H1c): Intraoral camera-assisted education reduces plaque accumulation on first permanent molars.

For this purpose, the study is planned as a randomized controlled trial with two groups: an intervention group and a control group. Data will be collected before the education and at the 1-month follow-up after the education to compare changes over time. A two-factor repeated measures ANOVA will be used to evaluate the differences between the groups.

A priori power analysis (G*Power 3.1) showed that at least 34 participants (17 for each group) are needed to detect a medium effect (f = 0.25, α = 0.05, 80% power). To reduce the risk of sample loss, a total of 40 child-parent pairs will be included. These pairs will be randomly assigned to either the intraoral camera-assisted education group or the standard verbal education group.

Intervention group: Receives intraoral camera-assisted oral hygiene education. Dental findings such as plaque, caries, and gingival inflammation, as well as brushing techniques, are visualized in real time. Disclosing agents highlight plaque-covered areas, and brushing demonstrations on the child's teeth are individualized using the Modified Stillman and cross-brushing techniques. Parents and children receive visual feedback to reinforce oral hygiene education.

Control group: Receives standard verbal oral hygiene education using a brushing model. The Modified Stillman and cross-brushing techniques are demonstrated verbally and on the model, without intraoral camera visualization.

Primary outcomes are changes in children's Plaque Index (PI), Gingival Index (GI), ICDAS caries scores, and parents' oral health literacy assessed using the Turkish version of the Oral Health Literacy Assessment Task for Pediatric Dentistry (TOHLAT-P).

Secondary outcomes are the Occlusal Plaque Index (OPI) on first molars and the Parent-Child Satisfaction Survey evaluating the intraoral camera-assisted education. Assessments will be conducted at baseline and 1-month follow-up, except for the satisfaction survey, which will be administered only at the 1-month follow-up. The study assesses whether visualized instruction provides additional benefits over verbal education alone in improving objective clinical measures and parental understanding, supporting enhanced preventive care in pediatric dental practice.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy children
* Age between 5-7 years, with at least one first permanent molar in the eruption stage
* No urgent treatment needs (e.g., dental trauma or pain)
* Voluntary participation with signed and verbal informed consent from parents, and willingness to attend follow-up visits regularly

Exclusion Criteria:

* Children with special healthcare needs, intellectual disabilities, or autism spectrum disorder
* Children with a Frankl Behavior Rating Scale score of 1 (Definitely negative)

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Children's Plaque Index (PI) | Baseline
  Plaque levels on the mesial, distal, buccal, and lingual surfaces of all present teeth, excluding partially erupted teeth, were assessed using the Silness and Löe Plaque Index (scores 0-3).
  Plaque Index and Criteria:
  0.Absence of microbial plaque
  1. Thin film of microbial plaque along the free gingival margin
  2. Moderate accumulation with plaque in the sulcus
  3. Large amount of plaque in sulcus or pocket along the free gingival margin
Children's Plaque Index (PI) | 1 month after intervention
  Plaque levels on the mesial, distal, buccal, and lingual surfaces of all present teeth, excluding partially erupted teeth, were assessed using the Silness and Löe Plaque Index (scores 0-3).
  Plaque Index and Criteria:
  0. Absence of microbial plaque
  1. Thin film of microbial plaque along the free gingival margin
  2. Moderate accumulation with plaque in the sulcus
  3. Large amount of plaque in sulcus or pocket along the free gingival margin
Children's Gingival Index (GI) | Baseline
  Gingival status was assessed on the mesial, distal, buccal, and lingual surfaces of all present teeth, excluding partially erupted teeth, using the Löe and Silness Gingival Index (0-3).
  Gingival Index (GI) and Criteria:
  0. Normal gingiva; no inflammation; no discoloration (erythema); no bleeding.
  1. Mild inflammation; slight erythema; minimal superficial alterations; no bleeding.
  2. Moderate inflammation; erythema; bleeding on probing.
  3. Severe inflammation; severe erythema and swelling; tendency to spontaneous bleeding; possible ulceration.
Children's Gingival Index (GI) | 1 month after intervention
  Gingival status was assessed on the mesial, distal, buccal, and lingual surfaces of all present teeth, excluding partially erupted teeth, using the Löe and Silness Gingival Index (0-3).
  Gingival Index (GI) and Criteria:
  0. Normal gingiva; no inflammation; no discoloration (erythema); no bleeding.
  1. Mild inflammation; slight erythema; minimal superficial alterations; no bleeding.
  2. Moderate inflammation; erythema; bleeding on probing.
  3. Severe inflammation; severe erythema and swelling; tendency to spontaneous bleeding; possible ulceration.
ICDAS Caries Score | Baseline
  Caries status of all present teeth, excluding partially erupted teeth, was recorded using the International Caries Detection and Assessment System (ICDAS).
  ICDAS Codes (International Caries Detection and Assessment System)
  0. Sound tooth surface
  1. First visual change in enamel
  2. Distinct visual change in enamel
  3. Localized enamel breakdown due to caries with no visible dentin
  4. Underlying dark shadow from dentin (with or without enamel breakdown)
  5. Distinct cavity with visible dentin
  6. Extensive distinct cavity with visible dentin
ICDAS Caries Score | 1 month after intervention
  Caries status of all present teeth, excluding partially erupted teeth, was recorded using the International Caries Detection and Assessment System (ICDAS).
  ICDAS Codes (International Caries Detection and Assessment System)
  0. Sound tooth surface
  1. First visual change in enamel
  2. Distinct visual change in enamel
  3. Localized enamel breakdown due to caries with no visible dentin
  4. Underlying dark shadow from dentin (with or without enamel breakdown)
  5. Distinct cavity with visible dentin
  6. Extensive distinct cavity with visible dentin
Parental Oral Health Literacy (TOHLAT-P) | Baseline
  Parents' oral health literacy, understanding of preventive care, and ability to support children's oral hygiene, assessed by TOHLAT-P.
  This questionnaire is used to assess parents' oral health knowledge. It measures three types of knowledge (factual, procedural, and conceptual) and includes cognitive process levels (remembering, understanding, and analyzing). The tool also uses literacy and numeracy skills. It has three sections.
  The maximum score for each section is 12, 26, and 14. The total score range is 0-52. Higher scores indicate higher oral health literacy.
Parental Oral Health Literacy (TOHLAT-P) | 1 month after intervention
  Parents' oral health literacy, understanding of preventive care, and ability to support children's oral hygiene, assessed by TOHLAT-P.
  This questionnaire is used to assess parents' oral health knowledge. It measures three types of knowledge (factual, procedural, and conceptual) and includes cognitive process levels (remembering, understanding, and analyzing). The tool also uses literacy and numeracy skills. It has three sections.
  The maximum score for each section is 12, 26, and 14. The total score range is 0-52. Higher scores indicate higher oral health literacy.

SECONDARY OUTCOMES:
Occlusal Plaque Index (OPI) | Baseline
  Plaque accumulation on the occlusal surfaces of permanent first molars will be assessed after plaque disclosure using an intraoral camera. The images will be analyzed with ImageJ software (National Institutes of Health, USA) by manually outlining the total occlusal surface area and the plaque-covered areas. All measurements will be performed by the same examiner and repeated at two different time points to reduce measurement error. Intra-examiner reliability will be evaluated using the intraclass correlation coefficient (ICC), and the occlusal plaque index (OPI) will be calculated as the percentage of plaque-covered area relative to the total occlusal surface area using the formula: OPI = (Plaque area / Occlusal surface area) × 100.
Occlusal Plaque Index (OPI) | 1 month after intervention
  Plaque accumulation on the occlusal surfaces of permanent first molars will be assessed after plaque disclosure using an intraoral camera. The images will be analyzed with ImageJ software (National Institutes of Health, USA) by manually outlining the total occlusal surface area and the plaque-covered areas. All measurements will be performed by the same examiner and repeated at two different time points to reduce measurement error. Intra-examiner reliability will be evaluated using the intraclass correlation coefficient (ICC), and the occlusal plaque index (OPI) will be calculated as the percentage of plaque-covered area relative to the total occlusal surface area using the formula: OPI = (Plaque area / Occlusal surface area) × 100.
Parent and Child Satisfaction with Intraoral Camera-Assisted Education | At 1 month after intervention
  In this study, children and parents will complete two short questionnaires to assess their perceptions of the use of an intraoral camera during dental examination. Responses will be recorded using a 5-point Likert-type scale ranging from strongly agree to strongly disagree, with higher scores indicating more positive perceptions of intraoral camera use.
  Child questionnaire
  1. I liked having photographs of my teeth taken with the intraoral camera.
  2. I felt comfortable while photographs of my teeth were taken using the intraoral camera.
  3. I would tell my friends about having my teeth photographed with an intraoral camera.
  Parent questionnaire
  1. The use of an intraoral camera helped us better understand dental treatment and oral hygiene instructions.
  2. The use of an intraoral camera improved our overall dental examination experience.
  3. I would recommend the use of an intraoral camera during dental examination to others.

CONTACTS AND LOCATIONS:
Overall Officials: Melis AKYILDIZ, Principal Investigator — Aydın Adnan Menderes University, Faculty of Dentistry
Locations (1):
- Aydın Adnan Menderes University, Faculty of Dentistry, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buldur B, Oguz E. Reliability and validity of the Turkish version of the Oral Health Literacy Assessment Task: Pathways between parental oral health literacy and oral health consequences in children. Int J Paediatr Dent. 2023 Mar;33(2):101-112. doi: 10.1111/ipd.13025. Epub 2022 Jul 26. PMID 35851730
- [Background] Carvalho JC. Chapter 9.2: Non-Operative Treatment of Coronal Caries. Monogr Oral Sci. 2023;31:149-171. doi: 10.1159/000530589. Epub 2023 Jun 26. PMID 37364559
- [Background] Duman, S., & Duruk, G. (2018). 6-12 Yaş Grubu Çocuklarda Daimi Birinci Büyük Azı Dişlerin Önemi ve Değerlendirilmesi - Derleme. Atatürk Üniversitesi Diş Hekimliği Fakültesi Dergisi, 28(4), 610-624.
- [Background] Gugnani N, Pandit IK, Srivastava N, Gupta M, Sharma M. International Caries Detection and Assessment System (ICDAS): A New Concept. Int J Clin Pediatr Dent. 2011 May-Aug;4(2):93-100. doi: 10.5005/jp-journals-10005-1089. Epub 2010 Apr 15. PMID 27672245
- [Background] Khan AA. The permanent first molar as an indicator for predicting caries activity. Int Dent J. 1994 Dec;44(6):623-7. PMID 7851995
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Murrell M, Marchini L, Blanchette D, Ashida S. Intraoral Camera Use in a Dental School Clinic: Evaluations by Faculty, Students, and Patients. J Dent Educ. 2019 Nov;83(11):1339-1344. doi: 10.21815/JDE.019.140. Epub 2019 Aug 12. PMID 31406005
- [Background] Nourallah AW, Splieth CH. Efficacy of occlusal plaque removal in erupting molars: a comparison of an electric toothbrush and the cross-toothbrushing technique. Caries Res. 2004 Mar-Apr;38(2):91-4. doi: 10.1159/000075931. PMID 14767164
- [Background] Ozgul BM, Sakaryali D, Senirkentli GB, Tirali RE, Cehreli SB. Do really parents brush their children's teeth better? Eur J Paediatr Dent. 2019 Dec;20(4):325-329. doi: 10.23804/ejpd.2019.20.04.13. PMID 31850778
- [Background] Pentapati KC, Siddiq H. Clinical applications of intraoral camera to increase patient compliance - current perspectives. Clin Cosmet Investig Dent. 2019 Aug 23;11:267-278. doi: 10.2147/CCIDE.S192847. eCollection 2019. PMID 31692486
- [Background] Schiller C, Ho H, Sobue T, Katechia B, Tadinada A. Value of an Intraoral Camera in Evaluating Restorations and Plaque in a Simulated Environment: Observational Experiences of Dentists in Pediatric Contexts to Establish a Proof of Concept. Cureus. 2024 Oct 21;16(10):e72012. doi: 10.7759/cureus.72012. eCollection 2024 Oct. PMID 39569297
- [Background] Schulz-Weidner N, Gruber M, Schraml EM, Wostmann B, Kramer N, Schlenz MA. Improving the Communication of Dental Findings in Pediatric Dentistry by Using Intraoral Scans as a Visual Aid: A Randomized Clinical Trial. Dent J (Basel). 2024 Jan 17;12(1):15. doi: 10.3390/dj12010015. PMID 38248223
- [Background] Sharma S, Yeluri R, Jain AA, Munshi AK. Effect of toothbrush grip on plaque removal during manual toothbrushing in children. J Oral Sci. 2012;54(2):183-90. doi: 10.2334/josnusd.54.183. PMID 22790411
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Tan WK, Chua DR. Parental use and acceptance of an accessible, commercially available intraoral camera for teledentistry in their children. Eur Arch Paediatr Dent. 2024 Apr;25(2):237-246. doi: 10.1007/s40368-024-00878-7. Epub 2024 Apr 21. PMID 38643420
- [Background] Wong HM, Bridges SM, Yiu CK, McGrath CP, Au TK, Parthasarathy DS. Validation of the Hong Kong Oral Health Literacy Assessment Task for paediatric dentistry (HKOHLAT-P). Int J Paediatr Dent. 2013 Sep;23(5):366-75. doi: 10.1111/ipd.12021. Epub 2013 Jan 24. PMID 23947421
- [Background] Yao Y, Luo A, Hao Y. Selective versus stepwise removal of deep carious lesions: A meta-analysis of randomized controlled trials. J Dent Sci. 2023 Jan;18(1):17-26. doi: 10.1016/j.jds.2022.07.021. Epub 2022 Aug 21. PMID 36643250
- [Background] Zouashkiani, T., & Mirzakhan, T. (2006). Parental Knowledge about Presence of the First Permanent Molar and Its Effect on Health of the Tooth in 7-8 Years Old Children. J Mashad Dent Sch, 30, 225-32.
- See also: This article introduces ICDAS, a standardized visual and clinical method for detecting and assessing dental caries from early to advanced stages, widely used in pediatric dentistry for accurate and early caries identification. — https://doi.org/10.5005/jp-journals-10005-1089
- See also: This study compared plaque removal efficacy of conventional and silicone toothbrushes in children aged 5-7, showing both methods were effective. — https://doi.org/10.23804/ejpd.2019.20.04.13